CLINICAL TRIAL: NCT06811766
Title: Comparative Effects of Strain-counterstrain and Muscle Energy Techniques on Neck Pain and Functional Disability in Patients with Cervicogenic Headache
Acronym: SCS METs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Kinza Fatima, Kfatima, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUFkinza
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Cervicogenic Headache
Keywords: CGH; SCS; METs
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: There will be two groups. Each group will receive different treatment techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Active Comparator): This group containing 27 participants
  Interventions: Other: Strain-counterstrain
- 2 (Active Comparator): This group also containing 27 participants
  Interventions: Other: Muscle energy techniques

INTERVENTIONS:
Other: Strain-counterstrain — This is a technique that uses gentle body positioning passively to treat muscles and joints pain. So, this can be effective for neck pain in patients with CGH
  Other Names: SCS
  Arms: 1
Other: Muscle energy techniques — This technique uses patient's own muscles to treat muscles and joint restrictions. So, this technique can be prove affective for neck pain and limited range in patients with CGH
  Other Names: METs
  Arms: 2

SUMMARY:
The primary objective of this study is to compare effects of SCS and METs on reduction of neck pain intensity and improvement in functional disability in individuals with CGH. The secondary objective is to assess the impact of both techniques on ROM in cervical spine

ELIGIBILITY:
Inclusion Criteria:

* participants who fulfill the criteria of international headache society.

Exclusion Criteria:

* participants who have cervicogenic headache after cervical injury or head surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 3 weeks
  To check pain intensity
Neck disability index | 3 weeks
  To check functional disability

SECONDARY OUTCOMES:
Goniometer | 3 weeks
  To measure range of motion